CLINICAL TRIAL: NCT01496820
Title: Effect of GO2KA1(Chitosan Oligosaccharide) on Postprandial Blood Glucose in Korean Adults: a Clinical Randomized Trial
Brief Title: A Randomized Trial to Assess the Efficacy and Safety of GO2KA1(Chitosan Oligosaccharide)on Blood Glucose Control
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KPB-HG-COS
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Impaired Fasting Glucose, Newly-diagnosed Type 2 Diabetes
MeSH Terms: interventions — GO2KA1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GO2KA1 (Experimental)
  Interventions: Dietary Supplement: GO2KA1
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GO2KA1 — GO2KA1(chitosan oligosaccharide)1500mg/day for 12weeks
  Arms: GO2KA1
Dietary Supplement: Placebo — placebo 1500mg/day for 12weeks
  Arms: Placebo

SUMMARY:
The effects of chitosan on blood glucose levels have been contradicting. Hypoglycemic effects of high molecular weight chitosan are related to diabetic models with hypoinsulinemia but have shown little effect on the blood glucose levels in hyperinsulinemia related diabetic models. Based on previous reports, high molecular weight chitosan either directly or indirectly related to insulin secretion in pancreas but has little effect on insulin resistance. In the present study, the effect of GO2KA1 (low molecular weight chitosan oligosaccharide) on blood glucose levels in Korean pre-diabetic adults, will be evaluated. The changes in postprandial blood glucose levels will be investigated in subjects with impaired fasting glucose or glucose tolerance.

DETAILED DESCRIPTION:
In the detailed description we believe that it will be wise to discuss about the long-term study of the effect of GO2KA1(Chitosan oligosaccharide: oligosaccharides derived from chitosan) on pre-diabetic individuals (in addition to the postprandial blood glucose levels). In the present study, we will investigate the effects of GO2KA1 on the level of postprandial blood glucose in adult Koreans with impaired fasting glucose or impaired glucose tolerance. Postprandial blood glucose levels will be tested for 2 hours at every 30 min interval after 75g-OGTT and the experimental group will be pre-fed with 500 mg of GO2KA1. Primary outcomes will be included change in HbA1c, insulin, glycemic AUC, and lipids(total cholesterol, triglyceride, and HDL).

This clinical study will be conducted with 60 subjects after explanation and accommodation about experimental protocols and model. To test under same condition, smoking and drinking water will be completely prohibit from 1 hour before and during the experiment. At first day, control experiment will be conducted without oral take of GO2KA1 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* males and females 20-75 years old
* impaired fasting glucose (FPG 100~125 mg/dL) or impaired glucose tolerance (PPG-2h 140~200 mg/dL)
* able to give informed consent

Exclusion Criteria:

* having received a diagnosis of diabetes or receiving treatment for diabetes
* having a history of ischemic heart disease, stroke, liver cirrhosis, chronic pancreatitis, pituitary disease, thyroid disease, adrenal gland disease, mental illness, gastrectomy, or advanced malignant tumor
* receiving corticosteroid or thyroid hormone medication
* being judged by the responsible physician of the local study center as unfit to participate in the study
* abnormal liver or kidney function tests (ALT or AST > 2 times the upper limit of normal
* elevated creatinine, males > 125 umol/L, females > 110 umol/L)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose(PPG) | Change from baseline in PPG at 12 weeks
  Primary outcome will be tested for 2 hours at every 30 min interval after 75g-OGTT and the experimental group will be pre-fed with 500 mg of GO2KA1.

SECONDARY OUTCOMES:
HbA1c | Change from baseline in HbA1c at 12 weeks
Insulin | Change from baseline in insulin at 12 weeks
glycemic AUC | Change from baseline in glycemic AUC at 12 weeks
Total cholesterol | Change from baseline in Total cholesterol at 12 weeks
Triglyceride | Change from baseline in triglyceride at 12 weeks
HDL-cholesterol | Change from baseline in HDL-cholesterol at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea